CLINICAL TRIAL: NCT00618397
Title: Phase I Trial to Determine Steady State Pharmacokinetics and Sedative Effects of Low Dose Ketamine Infusion
Brief Title: Pharmacokinetics of Low Dose Ketamine Infusion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitement
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Cindy Darnell, Assisant Professor Pediatrics, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 042006035
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Sedation; Opioid Tolerance
Keywords: ketamine; pharmacokinetics; sedation; critical care; opioid tolerance; NMDA Antagonist
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Ketamine will be administered in doses of 0.01mg/kg/hr, 0.1mg/kg/hr and 0.5mg/kg/hr to in PICU patients that meet eligibility criteria.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine administered in doses of 0.01mg/kg/hr, 0.1mg/kg/hr and 0.5mg/kg/hr to PICU patients.
  Other Names: Brand Name - ketalar

SUMMARY:
Opioids, such as fentanyl, are commonly used in PICU patients to provide comfort and pain control. Opioid tolerance, the need to increase the dose of medication to achieve the same effect,is seen in PICU children who require opioid infusions. Animals and human studies have shown that activation of the N-methyl-D-aspartate (NMDA) receptor is involved in the development of opioid tolerance and that deactivation of this receptor can slow the development of tolerance. Ketamine, an NMDA receptor antagonists, turns off the NMDA receptor. Ketamine is used to provide sedation and anesthesia in children. Its use in inhibiting the development of opioid tolerance has not been tested in children. We aim to determine ketamine's effectiveness in the treatment of tolerance in PICU patients who require fentanyl infusions to treat pain and discomfort .

Some physicians have reported using ketamine doses of 0.04mg/kg/hr to 0.5mg/kg/hr to inhibit opioid tolerance. We propose to study the sedative effect, and the metabolism of, three doses of ketamine, 0.1mg/kg/hr, 0.3mg/kg/hr, and 0.5mg/kg/hr.

Patients admitted to the PICU, requiring a breathing machine and fentanyl infusion for discomfort or pain control will be enrolled. Patients' age three to eighteen years will be enrolled. Patients will receive a ketamine infusion once their COMFORT scores indicate an adequate sedation/comfort level on their current sedation regimen. The COMFORT score is a validated scale that measures distress in PICU patients. The COMFORT score will be continued for the twelve hours the patient receives the ketamine to test whether the ketamine adds to the level of sedation. Blood samples during and following the ketamine infusion will be taken to determine how ketamine and norketamine (one of ketamine's metabolites) are used in the body.

To determine the effect of ketamine on tolerance it must be a ketamine dose that does not cause additional sedation. The goal of this study is to define a non-sedating dose of ketamine and define how it is used by the body. A non-sedating ketamine dose could be added to current sedation regimens allowing us to monitor the development of tolerance without the confusion of added sedation. The data obtained in this study will be used to design a study to further investigate the effect of ketamine on opioid tolerance.

DETAILED DESCRIPTION:
Background:

There has been an increasing awareness of the need for adequate sedation and analgesia in critically ill pediatric patients. The choices of treatment for pain are numerous, but in the Pediatric ICU parenteral opioids are most commonly used. At equipotent doses, all mu agonist opioids (morphine, fentanyl, meperidine and codeine) produce similar physiologic effects and side effects. Opioids can cause hypoventilation, hypotension, constipation, and may cause urinary retention. Patients receiving continuous opioid infusions experience not only these physiologic side effects, but also the side effects of dependence, tolerance and withdrawal. These lastly named side effects often complicate medical issues and contribute to longer ICU admissions.

There are numerous articles addressing the problem of opioid tolerance, dependence, and withdrawal . Despite repeated efforts, the mechanism of tolerance remains unclear. Current in-vitro and in-vivo investigations focus on five theories of opioid tolerance: receptor down-regulation, desensitization, internalization, alternative coupling, and functional antagonism. Recent studies suggest that receptor down-regulation is not the main mechanism in-vivo. Desensitization by receptor decoupling, receptor internalization and increased alternative coupling to stimulatory G-proteins have been demonstrated to be clinically insignificant. However, functional antagonism of the opioid effects seems to be clinically most important. This functional antagonism is mediated by the activation of N-methyl-D-aspartate (NMDA) receptors, up-regulation of adenylyl cyclase and nitric oxide synthase . Drugs blocking these mechanisms are promising in the treatment of opioid tolerance. Numerous in-vivo studies have focused on blocking the NMDA receptor. Studies in animals have shown a decrease in the development of opioid tolerance when NMDA antagonists are used . This effect has been escalated to the next level of investigation as several adult case reports and randomized controlled trials demonstrate patients receiving small, sub-anesthetic doses of ketamine respond with a subsequent dramatic decrease in opioid requirement. The doses of ketamine used in these case reports vary, from 1mg/kg/24 hours (0.04mg/kg/hr), to 0.1mg/kg/hr . Bell recently reviewed four randomized controlled trials in cancer patients receiving ketamine as an adjuvant to opioids for pain. Dosing and route of ketamine varied between trials. He cautiously concluded that there is promise in the potential efficacy of ketamine as an adjuvant to opioids for cancer pain . Another review reported that coadministration of ketamine reduced pain, analgesic consumption, and in some studies both . Suresh and Anand anecdotally report using 0.2mg/kg/hr-0.5mg/kg/hr in children with a resultant decreased need to escalate morphine infusion rates.

Part of the difficulty in determining an appropriate pediatric dose is the lack of clinical studies evaluating ketamine as adjuvant to opioids in children. There have been numerous attempts in adults to evaluate the effect of adding ketamine to opioids to improve pain management. Many of these studies were reviewed by Subraminiam. Of the fifty-seven studies reviewed, only seven used continuous infusion IV ketamine in addition to opioids. Of these seven studies, four reported significantly improved analgesia with the addition of ketamine. Of the fifty-seven studies, only four evaluated ketamine as an adjuvant to opioids in children. All of these studies were evaluating postoperative pain control and only one used continuous infusion ketamine. Of the four only one, evaluating preoperative ketamine administration, showed improvement in pain control .

In the future, we anticipate conducting a randomized, blinded, placebo controlled trial to evaluate the effect of low dose ketamine on the development of opioid tolerance. However, there is no standardized dose of ketamine for this role. The goal of this phase I trial to is to establish a dose of continuous infusion ketamine to be used in future studies, and to further the pharmacokinetic details of ketamine as a continuous infusion at this dose. There is currently no data describing the pharmacokinetics of low dose ketamine in children. These details would include plasma concentration, elimination rate, and half-life of ketamine and its primary metabolite norketamine. In addition to expanding the available data on ketamine this information could be useful in future studies. It has been reported that ketamine causes sedation in children at serum levels of 1 to 1.5 ug/ml, and that at levels less than 0.5ug/ml there are no sedative effects . The assumption can be made that at levels less than 1ug/ml ketamine is non-sedating, but this has not been tested.

While opioids are considered an analgesic, they also have sedative properties and are often the first-line drug for sedation in Pediatric ICU's even when true analgesia is not required . Fentanyl is frequently used in the Pediatric ICU at Children's Medical Center Dallas for the sedation/analgesia of patients requiring mechanical ventilation. A future study would use percent increase in fentanyl dose as a measure of tolerance. Patients would receive ketamine or placebo, in addition to the fentanyl infusion that is the standard of care for sedation in the Pediatric ICU. The fentanyl infusion would be titrated as per standard of care, with the addition of midazolam at the discretion of the primary team, to maintain adequate sedation. As tolerance develops there should be an increase in the fentanyl dose to maintain the same clinical effect. If ketamine does inhibit the development of tolerance then the ketamine group should remain adequately sedated with a smaller percent increase in fentanyl. For sedation to be a valid measure in this circumstance it would have to be known that the ketamine dose used was itself non-sedating.

The purpose of this study is to determine the sedative properties, and pharmacokinetics, of several low dose ketamine regimens. By determining the sedative profile of ketamine at these doses, we will be able to accurately define low dose ketamine as a dose that is nonsedating.

Hypothesis:

In PICU patients, age 3 years to 18 years receiving continuous fentanyl infusions and/or benzodiazepine infusions for mechanical ventilation, low dose ketamine will not cause an increase in sedation from baseline.

Study Design:

This will be a phase I trial evaluating ketamine at various doses for pharmacokinetics and the effect of over-sedation (sedation increased significantly from baseline defined as a six point change) according to the COMFORT score. The COMFORT score is an objective scale developed to measure distress in pediatric critical care patients . Its use in predicting optimal sedation for mechanically ventilated patients has been validated .

We will enroll patients admitted to the Pediatric Intensive Care Unit at Children's Medical Center Dallas for respiratory failure requiring intubation and mechanical ventilation. The PICU at Children's Medical Center is a 44 bed ICU that admits patients with a wide range of medical problems. In 2005 there were 118 patients admitted with the primary diagnoses of respiratory failure. Another 147 patients had secondary diagnoses of respiratory failure. We anticipate enrolling 15 patients over the course of one year.

Once patients are enrolled, the COMFORT score will be administered by nursing staff every four hours. When the patient has had scores of seventeen to twenty-six on two successive occasions, with no need for alteration of sedation regimen, they will be considered optimally sedated. At this time a ketamine infusion will be initiated per standard infusion pump. Ketamine will be administered as an infusion for twelve hours. The ketamine doses to be administered are within the dosage range of ketamine used in prior literature. It is felt that these doses are non-sedating. The first five patients enrolled in will receive ketamine at 0.01mg/kg/hr. The COMFORT score will continue to be administered every four hours for the twelve hours while the patient receives the ketamine infusion. If the COMFORT score is less than seventeen, the patient is considered over-sedated, and medication adjustments will be made by the primary team. The ketamine infusion will continue but the fentanyl and/or midazolam dose will be adjusted according to the primary care team. If the COMFORT score is more than twenty-six, the patient is considered under-sedated and will require medication adjustments. The ketamine infusion will not be changed but the fentanyl and or midazolam will be adjusted according to the primary care team. The COMFORT score will be repeated one hour after all medication changes.

If the COMFORT score is consistent with optimal sedation no medication changes will be made. If, in the opinion of the primary team, the patients requires a level of sedation resulting in a COMFORT score lower than 17 that patient will be removed from the study. Any patient who requires a change in the fentanyl or midazolam infusion will be removed from the study. If possible the ketamine infusion will be completed and serum levels drawn but the patient will not be included in the sedation portion of the study.

Prior to enrolling patients at the next dose, we will ensure that all serum levels are less than 1ug/ml. If levels are satisfactory, enrollment will begin at the next dose. The doses to be studied are 0.01mg/kg/hr, 0.1mg/kg/hr, and 0.5mg/kg/hr.

By enrolling five patients at each dose, we will be able to accurately define the pharmacokinetics as well as the sedation profile for each. In order to determine the pharmacokinetics of ketamine, blood samples to determine the serum concentration of ketamine and its primary metabolite, norketamine will be obtained. Whole blood samples of 400ul will be obtained via available venous or arterial catheter. If no catheter is available then the blood may be obtained via heel stick per current PICU standards. Serum samples will be obtained just prior to starting the ketamine infusion, six hours after starting the infusion, and at twelve hours after starting the infusion. Three additional samples will be obtained at two, four, and six hours after discontinuing the infusion. Assuming a one compartment open model and first order elimination the following parameters will be estimated: Plasma concentration, volume of distribution, elimination rate, half-life, dose and steady state concentration. The elimination half-life will be determined from the slope of the best-fit concentration versus time plot following discontinuation of the ketamine infusion. Ketamine and norketamine will be analyzed using a qualified LC-MS/MS method .

Throughout the study, patients will be monitored for adverse events. Should the patient develop any adverse events not related to their current medical condition including but not limited to nausea, vomiting, hypotension, hypertension, tachycardia, tremulousness, increased tone in extremities, seizures, cardiac arrhythmias, and/or hallucinations that can not be otherwise explained by the current medical condition, the ketamine infusion will be discontinued. Serum samples for elimination half-life will be obtained at two, four and six hours after discontinuing the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they meet the following criteria:
* Children age one three (3) years to eighteen (18) years, requiring admission to the Pediatric ICU, who require intubation for respiratory failure and continuous infusion fentanyl.
* Patients of both genders, all races and ethnic backgrounds will be eligible.
* Patients will need to have AST and ALT evaluated within the two weeks prior to enrollment, with the result being within two times the normal range. Patients who have not had AST and ALT evaluated within two weeks will have to be evaluated prior to enrollment. Serum will be evaluated for AST and ALT when convenient to other lab testing prior to enrollment.
* Patients meeting the above criteria will be eligible regardless of nutritional status, performance status or recovery from prior medical treatment.
* Patients will not be excluded if they require simultaneous infusions of sedation with benzodiazepine.
* Enrollment will require parental consent.

Exclusion Criteria:

* Patients will not be eligible if they meet any of the following criteria:
* Patients who are currently on oral analgesia or sedation
* Patients who have a prior history of drug or alcohol dependence/abuse.
* Patients who are allergic to opioids.
* Patients who are allergic to ketamine or any NMDA antagonist. Patients in whom significant elevation of blood pressure would constitute a serious hazard
* Patients with documented or clinical concern for elevated intracranial pressure.
* Patients with known liver dysfunction as evidenced by AST and ALT two times the normal limit within the past two weeks.
* Patients who are being medically paralyzed as part of their current treatment.
* Patients with any underlying neurologic condition, or impairment, which would interfere with their perception of, or response to, pain or discomfort.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To establish if continuous infusions of ketamine in doses of 0.01mg/kg/hr, 0.1mg/kg/hr and 0.5mg/kg/hr cause serum levels > 1 mcg/ml. | 6 and 12 hours after begining infusion

SECONDARY OUTCOMES:
To define the pharmacokinetics of continuous infusion ketamine in doses of 0.01mg/kg/hr, 0.1mg/kg/hr and 0.5mg/kg/hr. | 6 and 12 hours after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Darnell, MD, Principal Investigator — University of Texas
Locations (1):
- Children's Medical Center Dallas, University of Texas Southwestern, Dallas, Texas, United States